CLINICAL TRIAL: NCT03227068
Title: Nurse-Led Parent Educational Discharge Support Strategies (PEDSS) for Children Newly Diagnosed With Cancer
Brief Title: Parent Educational Discharge Support Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Children's Health System of Texas Children's Medical Center (Unknown); Cohen Children's Medical Center (Other); Levine Children's Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Maine Children's Cancer Program at Maine Medical Center (Unknown); Medical University of South Carolina Children's Hospital (Unknown); Nationwide Children's Hospital (Other); Northwestern Medicine Central DuPage Hospital (Unknown); St. Jude Children's Research Hospital (Other); St. Louis Children's Hospital (Other); St. Peter's University Hospital (Unknown); University of Wisconsin Health American Children's Hospital (Unknown); West Virginia Univeristy Medicine (Unknown); King Faisal Specialist Hospital & Research Center (Other); Nicklaus Children's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00077090
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Educational Activities
Keywords: pediatric oncology; parent

STUDY DESIGN:
Intervention Model Description: All subjects in both groups will receive education regarding their specific disease and treatment in accordance with current practices. Cancer care providers describe detailed side effects of treatment to parents during the treatment consent process. In addition, all parents will receive standard discharge education before hospital discharge including a list of home medications, and information regarding whom to call for emergencies. The PEDSS - symptom management and PEDSS - support for the caregiver are additional tools designed to reinforce care after the initial hospital discharge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEDSS - symptom management (Experimental): Content for the PEDSS - symptom management includes the most commonly experienced treatment-related physical symptoms, descriptions of each symptom, strategies to reduce symptom distress, and when and how to contact the cancer care team.
  Interventions: Other: PEDSS - symptom management
- PEDSS - support for the caregiver (Experimental): Content for the PEDSS - support for the caregiver includes five topics and suggestions on how caregivers can care for themselves during this time.
  Interventions: Other: PEDSS - support for the caregiver

INTERVENTIONS:
Other: PEDSS - symptom management — All subjects will receive education regarding their specific disease and treatment in accordance with current practices. Cancer care providers describe detailed side effects of treatment to parents during the treatment consent process. In addition, all parents will receive standard discharge education before hospital discharge, which includes a list of home medications and information regarding whom to call for emergencies. The PEDSS - symptom management will be delivered prior to the initial hospital discharge. The nurse will review the symptom management worksheet verbally with the parent, then distribute the written worksheet to the parent.
  Arms: PEDSS - symptom management
Other: PEDSS - support for the caregiver — All subjects will receive education regarding their specific disease and treatment in accordance with current practices. Cancer care providers describe detailed side effects of treatment to parents during the treatment consent process. In addition, all parents will receive standard discharge education before hospital discharge, which includes a list of home medications and information regarding whom to call for emergencies. The PEDSS - support for the caregiver will be delivered prior to the initial hospital discharge. The nurse will review the worksheet verbally with the parent, then distribute the written worksheet to the parent.
  Arms: PEDSS - support for the caregiver

SUMMARY:
After the initial hospitalization, parents of children newly diagnosed with cancer assume responsibility for assessing and managing their care; however, parents are often overwhelmed with information received throughout the hospitalization and are apprehensive about caring for their child at home. Parents want concise, focused information on how to care for their child after the hospital discharge. Two parent education discharge support strategies (PEDSS) were created to use at hospital discharge. PEDSS consists of a symptom management intervention and a support for the caregiver intervention. A cluster randomized control trial will assess the effectiveness and feasibility of the two different interventions.

DETAILED DESCRIPTION:
Providing education to parents of children newly diagnosed with cancer is a primary component of nursing practice, but best practices regarding delivery of information are not known. Parents often report confusion and worry with the complexity and large volume of information received during the initial hospitalization that leads to concerns in caring for their child after discharge. In addition, the amount and content of education is not standardized across institutions. This results in considerable variability in educational practices, including symptom education. During a recent qualitative study, parents described helpful discharge education strategies as having written materials, keeping information concise, and receiving anticipatory guidance so they knew what to expect. These preferences were succinctly summarized by a mother of a child newly diagnosed with leukemia who stated "…it would be nice to have one sheet of paper that just said 'these are the signs that you're looking for at home'." The purpose of this research study is to implement and evaluate parent educational discharge support strategies (PEDSS) for parents of children newly diagnosed with cancer. Findings from this study will provide a framework for nurses to deliver concise and consistent information to parents of children newly diagnosed with cancer, and will assist parents with their child after hospital discharge.

The goal of this study is to determine the effectiveness and feasibility of two parent education discharge support strategies (PEDSS - symptom management vs. PEDSS - support for the caregiver) for parents of children newly diagnosed with cancer. Specific aims of the study include:

Specific Aim 1: Explore the effects of parent education discharge support strategies on childhood cancer symptoms (fever, pain, fatigue, nausea, appetite changes, and sleep problems) and parents' perception of their ability to care for their child with a new cancer diagnosis during the first two months following the initial hospital discharge.

Specific Aim 2: Determine whether implementation of parent education discharge support strategies decreases unplanned utilization of healthcare services (unscheduled clinic visits, emergency room visits, unplanned hospitalizations), and preventable toxicity (malnutrition, sepsis) among children with cancer during the first two months following the initial hospitalization.

Specific Aim 3: Examine the feasibility and fidelity of implementing the PEDSS at the initial hospital discharge among parents of newly diagnosed children with cancer for use through the first two months following hospital discharge at participating Magnet institutions.

ELIGIBILITY:
Inclusion Criteria:

* A parent (referred to as "parent" but includes a parent or legal guardian) of a patient 3 to 17 years of age who is newly diagnosed with any type of malignant disease on an inpatient oncology unit
* Must speak English, Spanish, or Arabic
* Child will be or is receiving chemotherapy and/or radiation therapy

Exclusion Criteria:

* A parent of a child diagnosed with histiocytosis or any hematological disease considered non-malignant
* A parent whose child received the initial cancer diagnosis and initial cancer treatment while hospitalized on a non-oncology unit (i.e., surgical ward)
* A parent of a child who is experienced a relapse of a malignant disease
* A parent who is the primary caregiver of the child with cancer and is illiterate

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 289 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Change from baseline pain severity to two months | At baseline and monthly for two additional months
  Wong-Baker Faces Scale
Change from baseline fatigue severity to two months | At baseline and monthly for two additional months
  Categorized as none to mild or moderate to severe from the Adolescent Fatigue Scale for adolescents 13-17 years of age, the Childhood Fatigue Scale for children 7-12 years of age, or the Parent Fatigue Scale to obtain proxy responses from parents of children < 7 years of age
Change from baseline nausea severity to two months | At baseline and monthly for two additional months
  Visual Analogue Scale in the form of a thermometer that rates the severity of nausea from 0-100
Change from baseline appetite changes to two months | At baseline and monthly for two additional months
  Simplified Nutritional Appetite Questionnaire, 4-item asking about child's appetite and rated on a 5-point Likert Scale
Change from baseline sleep disturbances to two months | At baseline and monthly for two additional months
  The Sleep Wake Scale
Change from baseline pain behavior to two months | At baseline and monthly for two additional months
  PROMIS® Pediatric - Pain Behavior Short Form

SECONDARY OUTCOMES:
Change of baseline parents' perception of their ability to care for their child with a new cancer diagnosis to two months | At baseline and monthly for two additional months
  Seven items asking the parent to rate perceptions of the care of their child's symptoms on a 5-point Likert scale
Unplanned utilization of healthcare services | At one and two months from start of study
  Combined frequency of the number of unscheduled clinic visits, emergency room visits, and unplanned hospitalizations
Change in baseline nutritional status to two months | At baseline and monthly for two additional months
  Body mass index
Sepsis | At one and two months from start of study
  Frequency of septic events over the past month
PEDSS intervention feasibility | At baseline
  Nurse documentation of completion of PEDSS discussion and distribution of PEDSS worksheet
PEDSS intervention satisfaction | At two months after intervention delivery
  Descriptive items asking about timing of intervention and frequency of intervention use then 6 items scored on a 5-point Likert scale asking about ease of use and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Hockenberry, PhD, Principal Investigator — Duke University; Megan Arthur, BS, Study Director — Duke University
Locations (16):
- United States (15):
  - Nicklaus Children's Hospital, Miami, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Central DuPage Hospital, Winfield, Illinois
  - Maine Children's Cancer Program at Maine Medical Center, Scarborough, Maine
  - St. Louis Children's Hospital, St Louis, Missouri
  - St. Peter's University Hospital, New Brunswick, New Jersey
  - Cohen Children's Medical Center Northwell Health, New Hyde Park, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Medical University of South Carolina Children's Hospital, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Health System of Texas Children's Medical Center, Dallas, Texas
  - West Virginia University Medicine, Morgantown, West Virginia
  - University of Wisconsin Health American Children's Hospital, Madison, Wisconsin
- King Faisal Specialist Hospital and Research Centre-Riyadh, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Each site PI participating in the study will receive a copy of their anonymous data upon completion of the study.